CLINICAL TRIAL: NCT03232359
Title: Assessment of Immature Platelet Fraction in Pregnancy-Associated Thrombotic Microangiopathy
Brief Title: Immature Platelet Fraction as a Promising Biomarker in Prediction Outcome of HELLP Syndrome
Status: Completed | Type: Observational
Sponsor: AYMAN ABDELKADER MOHAMED ABDELKADER (Other)
Responsible Party: Sponsor-Investigator, AYMAN ABDELKADER MOHAMED ABDELKADER, doctor, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Other Study IDs: AAMABDELKADER 3
Record Dates: First submitted 2017-07-23; First posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Pre-Eclampsia, Severe; HELLP Syndrome; Microangiopathy
MeSH Terms: conditions — Pre-Eclampsia; HELLP Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SPE/HELLP group: This group included 24 pregnant women (gestational age of >20 weeks) who were diagnosed as having TMA with provisional diagnosis of pre-eclampsia, HELLP syndrome. immature platelets fraction assessment within 12 hours of diagnosis
  Interventions: Diagnostic Test: immature platelets fraction
- TTP/HUS group: This group included 13 pregnant women (gestational age of >20 weeks) who were diagnosed as having TMA with provisional diagnosis of TTP/HUS. HELLP syndrome. immature platelets fraction assessment within 12 hours of diagnosis
  Interventions: Diagnostic Test: immature platelets fraction
- Control group: This group included 20 pregnant women (gestational age of >20 weeks) having normal pregnancy with normal blood pressure and platelet count.
  Interventions: Diagnostic Test: immature platelets fraction

INTERVENTIONS:
Diagnostic Test: immature platelets fraction — IPF-% and A-IPC using a reticulocyte detection channel CBC auto analyzer

SUMMARY:
Immature platelet fraction is a non-invasive test of real time thrombopoiesis. High IPF% has been suggested as an indicator of thrombocytopenia due to rapid platelet consumption. IPF% is able to discriminate between patients with TTP/HUS or SPE/HELLP

DETAILED DESCRIPTION:
Thrombotic microangiopathy (TMA) syndromes are extraordinarily diverse. Thrombotic thrombocytopenic purpura (TTP) and hemolytic uremic syndrome (HUS) are the two most well known, and are considered to be the most serious. TTP-HUS occurs more commonly in women and among women is commonly associated with pregnancy.

Nevertheless, there are other pregnancy conditions that may manifest with TMA, including preeclampsia, eclampsia, HELLP syndrome (hemolysis, elevated liver enzymes, and low platelet count), in addition to acute fatty liver of pregnancy, antiphospholipid syndrome, and systemic lupus erythematosis.

Assessment of immature platelets was introduced as a non-invasive test of real time thrombopoiesis. They are newly released in the circulation with a larger size & greater RNA content than mature platelets, and can be measured by automated haematology analyzer equipped with reticulocyte detection channel and described as immature platelet fraction (%-IPF) and immature platelet count (A-IPC).

A high %-IPF has been suggested as an indicator of thrombocytopenia due to rapid platelet consumption, while a low %-IPF is characteristic of bone marrow suppression states. %-IPF/A-IPF has the competency to be performed routinely and, therefore, can provide therapeutic and diagnostic feedback in the life threatening conditions.

The present study aimed to show the utility of estimating %-IPF and A-IPC using a reticulocyte detection channel CBC autoanalyzer as a simple reproducible blood analysis to be employed in the differential diagnosis of pregnancy-associated thrombotic microangiopathic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Older than 20 years of age
* Pregnant with singleton intrauterine pregnancy
* More than 20 weeks of gestation

Exclusion Criteria:

* Congenital malformation and fetuses with chromosomal or genetic syndrome.
* Recent blood transfusion.
* Refusal to participate in the study.
* BMI <18.
* Placental abnormalities like velamentous insertion.
* Multiple pregnancies.
* Known kidney disease.
* History of auto immune disease.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: SPE/HELLP group. This group included 24 pregnant women (gestational age of >20 weeks) who were diagnosed as having TMA with provisional diagnosis of pre-eclampsia, HELLP syndrome.
  Group 2: TTP/HUS group. This group included 13 pregnant women (gestational age of >20 weeks) who were diagnosed as having TMA with provisional diagnosis of TTP/HUS.
  Group 3: Control group. This group included 20 pregnant women (gestational age of >20 weeks) having normal pregnancy with normal blood pressure and platelet count.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
clinical response after delivery | 48 hours after delivery
  clinical and laboratory changes after delivery

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2015-01-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03232359/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03232359/SAP_001.pdf